CLINICAL TRIAL: NCT05592418
Title: A Randomized, Double Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Ampligen® in Patients With Post-COVID Conditions
Brief Title: Study to Evaluate the Efficacy and Safety of Ampligen in Patients With Post-COVID Conditions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIM ImmunoTech Inc. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMP-518
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Post COVID-19 Condition; Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — poly(I).poly(c12,U); Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ampligen / rintatolimod (Experimental): Subjects will receive rintatolimod (intravenous [IV]), up to 400 mg twice weekly for 12 weeks.
  Interventions: Drug: Rintatolimod
- Placebo / Saline (Placebo Comparator): Subjects will receive placebo / normal saline (intravenous [IV]), up to 160 mL twice weekly for 12 weeks.
  Interventions: Other: Placebo / Normal Saline

INTERVENTIONS:
Drug: Rintatolimod — 100 to 400 mg twice weekly
  Other Names: Ampligen; poly I : poly C12U; Rintatolimod (poly I : poly C12U)
  Arms: Ampligen / rintatolimod
Other: Placebo / Normal Saline — 40 to 160 mL twice weekly
  Arms: Placebo / Saline

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Ampligen® administered twice weekly by intravenous (IV) infusions in subjects experiencing the Post-COVID Condition of fatigue.

DETAILED DESCRIPTION:
This is a Phase 2, two-arm, randomized, double blind, placebo controlled multicenter study to evaluate the efficacy and safety of Ampligen® in patients experiencing the Post-COVID Condition of fatigue. Patients will be randomized 1:1 to receive twice weekly IV infusions of Ampligen® or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult between 18 to 60 (inclusive) years of age at time of enrollment.
2. Prior confirmed COVID-19 diagnosis by standard RT-PCR assay or equivalent testing at least 12 weeks prior to baseline.

   Note: For subjects with COVID-19 symptoms who were not tested for the presence of SARS-CoV-2, a positive serum antibody test for SARS-CoV-2 will be sufficient in subjects not vaccinated for COVID-19 or it can be shown that the positive antibody cannot be associated with the COVID-19 vaccination.
3. Laboratory confirmed negative SARS-CoV-2 (COVID-19) infection by a government approved test / kit at time of enrollment.
4. Subject meets the criteria of fatigue per the 1994 CDC Case Definition for Chronic Fatigue Syndrome (CFS): Unexplained persistent or relapsing chronic fatigue that is of new or definite onset (i.e., not lifelong), is not the result of ongoing exertion, is not substantially alleviated by rest, and results in substantial reduction in previous levels of occupational, educational, social, or personal activities. The fatigue must have persisted or recurred during 3 or more consecutive months of illness and must not have preceded the onset of the COVID-19 symptoms.
5. PROMIS® Fatigue- Short Form 7a score of ≥21 at screening and baseline.
6. Electrocardiogram (ECG) with no clinically significant findings as assessed by the Investigator.

   Note: Below are the examples of clinically significant ECG abnormalities:
   * Previous documented evidence of myocardial infarction or recent significant change in the resting EKG suggesting infarction or other acute cardiac events.
   * Current symptoms of coronary insufficiency (i.e. - angina pectoris and/or ST segment depression on EKG).
   * Evidence of uncontrolled atrial or frequent or complex ventricular ectopy, or myocardial conduction defect which would increase the risk of syncope (for example, second degree or higher A-V block).
7. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.
8. Men and women of childbearing potential and their partner must agree to use two medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], or one of the following methods of birth control (intrauterine devices, bilateral tubal occlusion, or vasectomy) or must practice complete sexual abstinence for the duration of the study (excluding women who are not of childbearing potential and men who have been sterilized).
9. Females of child-bearing potential must have a negative urine pregnancy test at Screening Visit and prior to receiving the first dose of study drug; and Male participants must agree to use contraception and refrain from donating sperm for at least 90 days after the last dose of study intervention.
10. Subject is willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures and study restrictions.

Exclusion Criteria:

1. Inability to provide informed consent or to return to the Investigator's site for scheduled infusions and evaluations.
2. Exhibiting signs of moderate or severe pulmonary disease (such as COPD, asthma, or pulmonary fibrosis).
3. Ongoing requirement of oxygen therapy.
4. Pulse oxygen saturation (SpO2) of <94% on room air at the time of screening.
5. Thrombocytopenia (platelets <100×109/L), anemia (hemoglobin <9.0 g/dL), or leukopenia (WBC <3×109/L) on screening labs
6. History of splenectomy.
7. Known hypercoagulable state or at increased risk of thrombosis (e.g., due to immobility)
8. Liver cirrhosis or patient showing signs of clinical jaundice at the time of screening.
9. Transaminase (ALT or AST) >3X ULN or total bilirubin >2X ULN at screening
10. Chronic kidney disease stage 4 or requiring dialysis at the time of screening.
11. Estimated GFR <60 mL/min/1.73 m2 at the time of screening
12. NYHA Class III or IV congestive heart failure (CHF).
13. Exhibiting signs of uncontrolled hypo-or hyper-thyroidism at the time of Screening.
14. Diagnosis of autoimmune disease (e.g., SLE, rheumatoid arthritis, psoriasis) at the time of screening
15. Uncontrolled rheumatologic disorders at the time of screening.
16. Diagnosis of sleep apnea (central or obstructive) at the time of screening.
17. History of organ transplantation or are candidates for organ transplantation at the time of screening.
18. History of Chronic Fatigue Syndrome prior to COVID-19 infection.
19. History of fibromyalgia prior to COVID-19 infection.
20. History of major psychiatric disorder including psychotic or melancholic features, bipolar disorders, schizophrenia of any subtype, schizoaffective disorder, major depression delusional disorders of any subtype, dementias of any subtype, anorexia nervosa or bulimia nervosa.
21. Any malignancy within the past 5 years, excluding successfully treated basal cell carcinoma or squamous cell carcinoma without evidence of metastases.
22. Any other clinically significant serious systemic diseases, chronic or intercurrent active medical disorder and other reasons which would interfere with study conduct or study results interpretation per the Investigator.
23. Chronic or intercurrent acute medical disorder or disease making implementation or interpretation of the protocol or results difficult or unsafe per the investigator.
24. Therapy with interferons, interleukins, or other cytokines or investigational drugs within 6 weeks of beginning study medication. Subjects must give written informed consent prior to discontinuation of investigational drugs.
25. Treatment with any of the following therapies within the eight (8) weeks immediately preceding the start of study baseline or during baseline: systemic glucocorticoids (i.e., hydrocortisone, prednisone, etc.) or mineralocorticoids (i.e., fludrocortisone (Florinef), etc.), interferons, interleukin-2, systemic antivirals, gamma globulin or investigational drugs or experimental agents not yet approved for use in the United States.
26. Prior participation in an Ampligen® study.
27. Medical necessity, as determined by the patient's primary doctor or the principal investigator, to continue aspirin (ASA) or non-steroidal anti-inflammatory (NSAID) drugs for 20 consecutive days or for more than 10% of the study duration.
28. History of congestive heart failure, suspected or known dissecting aneurysm, recent systemic or pulmonary embolus or myocardial infarction (≤ 6 months), severe valvular heart disease, ventricular aneurysm, active or suspected myocarditis or pericarditis, thrombophlebitis or intracardiac thrombi, or acute infection.
29. Evidence of moderate or severe obstructive pulmonary disease.
30. Resting diastolic blood pressure > 115 mm Hg or resting systolic blood pressure > 200 mm Hg.
31. Uncontrolled metabolic disease (e.g., diabetes, thyrotoxicosis, or myxedema).
32. Concurrent use of any beta blockers and/or bronchodilators which cannot remain at a stable dosage level during baseline and the study.
33. History of alcohol or other substance abuse within two (2) years before the onset of acute COVID-19 or at any time afterward.
34. History of suicidal ideation, suicide attempt, or suicidal behavior within two (2) years of baseline. A score of 10 or greater on the PHQ-9 at Baseline indicates symptoms of depression and will exclude subject. A score of greater than zero on question nine (9) of the PHQ-9 at Baseline indicates suicidal ideation and will exclude subject.
35. Pregnant or breast feeding.
36. Participation in another study for an investigational treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Strayer, MD, Study Director — AIM ImmunoTech Inc.
Locations (5):
- United States (5):
  - Hope Clinical Research, Canoga Park, California
  - 310 Clinical Research, Inglewood, California
  - Acclaim Clinical Research, San Diego, California
  - Alfa Medical Research, Davie, Florida
  - Zenos Clinical Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 142 screened participants, 80 met inclusion criteria and were randomized to treatment.
Groups:
- Ampligen / Rintatolimod: Subjects received rintatolimod (intravenous [IV]), up to 400 mg twice weekly for 12 weeks.
  Rintatolimod: 100 to 400 mg twice weekly
- Placebo / Saline: Subjects received placebo / normal saline (intravenous [IV]), up to 160 mL twice weekly for 12 weeks.
  Placebo / Normal Saline: 40 to 160 mL twice weekly
Period: Overall Study
Arm/Group | Ampligen / Rintatolimod | Placebo / Saline
Started | 40 | 40
Completed | 36 | 30
Not Completed | 4 | 10
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 2 | 7

BASELINE CHARACTERISTICS:
Population: Total of 80 subjects were enrolled. Forty were randomized to each study group (Ampligen® or placebo). All subjects received at least one treatment.
Groups:
- Ampligen® /Rintatolimod: Subjects received rintatolimod (intravenous [IV]), up to 400 mg twice weekly for 12 weeks.
  Rintatolimod: 100 to 400 mg twice weekly
- Placebo/Saline: Subjects received placebo / normal saline (intravenous [IV]), up to 160 mL twice weekly for 12 weeks.
  Placebo / Normal Saline: 40 to 160 mL twice weekly
- Total: Total of all reporting groups
Arm/Group | Ampligen® /Rintatolimod | Placebo/Saline | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Adult between 18 to 60 (inclusive)years of age at time of enrollment
  years | 37.8 (11.03) | 34.8 (10.08) | 36.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 21 | 23 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Hispanic or Latino Not Hispanic or Latino
  Participants
    Hispanic or Latino | 30 | 24 | 54
    Not Hispanic or Latino | 10 | 16 | 26
    Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black or African American | 3 | 7 | 10
  White | 34 | 30 | 64
  Other | 2 | 2 | 4
Height (cm) [Mean (Standard Deviation); unit: cm] — At screening visit Height of subjects in cm were collected.
  cm | 169.5 (12.97) | 170.2 (10.15) | 169.9 (11.58)
Weight (kg) [Mean (Standard Deviation); unit: kg] — Weight of subjects in kg were collected.
  kg | 85.6 (20.95) | 87.8 (21.72) | 86.7 (21.23)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — BMI (kg/m^2) = Weight (kg)/[Height (cm)/100]^2
  kg/m^2 | 29.5 (5.91) | 30.3 (7.73) | 29.9 (6.85)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 13 in PROMIS Fatigue Score (T-Score)
Description: Change in mean fatigue T-score as measured by PROMIS® (Patient-Reported Outcomes Measurement Information System) Fatigue short form 7a that assess a range of self-reported symptoms, from mild subjective feelings of tiredness to extreme exhaustion. The lowest possible raw score is 7; the highest possible raw score is 35. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, with a standard deviation of 10 points. The lowest possible T-score is 29.4; the highest possible T-score is 83.2. A higher T-score represents more of the concept being measured, meaning the higher the T-Score, the worse the fatigue of the individual. Scores <55 are within normal limits, 55-60 mild, 61-70 moderate, and >70 severe fatigue.
Time Frame: Baseline and Week 13
Population: The Modified Intent-to-Treat (mITT) Population defined as the set of subjects who received at least one dose of study treatment (Ampligen® or placebo).
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Ampligen / Rintatolimod | Placebo / Saline
Number analyzed (Participants) | 40 | 40
T-Score
  Baseline | 69.9 (9.31) | 69.4 (7.51)
  change from Baseline at week 13: number analyzed (Participants) | 37 | 30
  change from Baseline at week 13 | -25.4 (11.2) | -25.8 (11.85)
Statistical Analysis 1: Comparison: Ampligen / Rintatolimod vs Placebo / Saline; Test type: Superiority; p = 0.9851, ANCOVA; Mean Difference (Final Values) = 0.0288, 95% CI 2-sided [-3.0397 to 3.0972] — LS Mean difference = LS Mean of Ampligen® - LS Mean of Placebo

2. Secondary Outcome: Change From Baseline to Week 6 in PROMIS Fatigue Score (T-Score)
Description: as for outcome 1
Time Frame: Baseline to Week 6
Population: The Modified Intent-to-Treat (mITT) population is defined as the set of subjects who have received at least one dose of study treatment (Ampligen® or placebo).
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Ampligen / Rintatolimod | Placebo / Saline
Number analyzed (Participants) | 40 | 40
T-Score
  Baseline | 69.9 (9.31) | 69.4 (7.51)
  change from baseline at week6-V12: number analyzed (Participants) | 35 | 33
  change from baseline at week6-V12 | -23.0 (13.65) | -19.6 (15.58)
Statistical Analysis 1: Comparison: Ampligen / Rintatolimod vs Placebo / Saline; Test type: Superiority; p = 0.3095, ANCOVA; Mean Difference (Final Values) = -1.9076, 95% CI 2-sided [-5.6279 to 1.8128]

3. Secondary Outcome: Change From Baseline to Week 13 in PROMIS Fatigue Score (T-Score), Excluding Response to Item Seven
Description: Change in mean fatigue T-score as measured by PROMIS® (Patient-Reported Outcomes Measurement Information System) Fatigue short form 7a that assess a range of self-reported symptoms, from mild subjective feelings of tiredness to extreme exhaustion. For this endpoint, the last question of "How often did you have enough energy to exercise strenuously" was excluded. Therefore, the lowest possible raw score is 6; the highest possible raw score is 30. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, with a standard deviation of 10 points. The lowest possible T-score is 33.4; the highest possible T-score is 76.8. A higher T-score represents more of the concept being measured, meaning the higher the T-Score, the worse the fatigue of the individual.
Time Frame: Baseline to Week 6 and 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Ampligen / Rintatolimod | Placebo / Saline
Number analyzed (Participants) | 40 | 40
T-Score
  Baseline | 66.2 (7.23) | 66.1 (5.98)
  change from baseline at Week6-V12: number analyzed (Participants) | 35 | 33
  change from baseline at Week6-V12 | -23.8 (14.16) | -20.8 (16.89)
  change from baseline at Week13-V26: number analyzed (Participants) | 37 | 30
  change from baseline at Week13-V26 | -27.1 (12.37) | -28.3 (12.32)
Statistical Analysis 1: Comparison: Ampligen / Rintatolimod vs Placebo / Saline; Test type: Superiority; p = 0.7663, ANCOVA; Mean Difference (Final Values) = 0.6086, 95% CI 2-sided [-3.4656 to 4.6829] — LS Mean difference = LS Mean of Ampligen® - LS Mean of Placebo

4. Secondary Outcome: Change From Baseline to Week 6 and Week 13 in Distance Traveled During 6-minute Walk Test (6MWT)
Description: The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance.
Time Frame: Baseline to week 6 and week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Ampligen® /Rintatolimod | Placebo/Saline
Number analyzed (Participants) | 40 | 40
Meters
  Baseline | 317.7 (79.85) | 312.1 (82.86)
  Change from baseline at week6-V12: number analyzed (Participants) | 37 | 34
  Change from baseline at week6-V12 | -2.1 (90.77) | 1.3 (87.64)
  Change from baseline at week13-V26: number analyzed (Participants) | 37 | 30
  Change from baseline at week13-V26 | 89.1 (108.18) | 69.3 (90.47)
Statistical Analysis 1: Comparison: Ampligen® /Rintatolimod vs Placebo/Saline; Test type: Superiority; p = 0.3162, ANCOVA; Mean Difference (Final Values) = 23.7749, 95% CI 2-sided [-23.2463 to 70.7962] — LS Mean difference = LS Mean of Ampligen® - LS Mean of Placebo

5. Secondary Outcome: Percentage of Subjects With Minimal Clinically Important Difference (MCID)
Description: Percentage of subjects with increase of at least 54 m from baseline in the Six-Minute Walk Test (6MWT) at the end of 12-week treatment phase presented and summarized descriptively by treatment group.
Time Frame: End of 12 week treatment phase
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ampligen / Rintatolimod | Placebo / Saline
Number analyzed (Participants) | 39 | 35
Participants | 39 | 35
Statistical Analysis 1: Comparison: Ampligen / Rintatolimod vs Placebo / Saline; P-value is from The Cochran-Mantel-Haenszel test (CMH) stratified by stratification factors; Test type: Superiority; Since all patients analyzed achieved MCID, there are no comparison results

6. Secondary Outcome: Change From Baseline to Week 6 and 13 in PROMIS Cognitive Function Converted Score (T-Score).
Description: Change in mean cognitive function T-score as measured by PROMIS® (Patient-Reported Outcomes Measurement Information System) Cognitive Function - Abilities short form 8a that assesses self-perceived cognitive deficits. The lowest possible raw score is 8; the highest possible raw score is 40. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, with a standard deviation of 10 points. The lowest possible T-score is 23.27; the highest possible T-score is 67.09. A higher T-score represents more of the concept being measured, meaning the higher the T-Score, the better the cognitive function of the individual. Scores >45 are within normal limits, 40-45 mild, 30-40 moderate, and <30 severe cognitive dysfunction.
Time Frame: Baseline to Week 6 and 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Ampligen / Rintatolimod | Placebo / Saline
Number analyzed (Participants) | 40 | 40
T-Score
  Baseline: number analyzed (Participants) | 37 | 39
  Baseline | 50.0 (11.67) | 46.3 (10.31)
  Change from Baseline to week6-V12: number analyzed (Participants) | 32 | 32
  Change from Baseline to week6-V12 | 5.5 (15.17) | 8.6 (15.16)
  Change from baseline to week13-V26: number analyzed (Participants) | 34 | 29
  Change from baseline to week13-V26 | 2.8 (18.63) | 8.0 (18.08)
Statistical Analysis 1: Comparison: Ampligen / Rintatolimod vs Placebo / Saline; Test type: Superiority; p = 0.4232, ANCOVA; Mean Difference (Final Values) = -3.2342, 95% CI 2-sided [-11.2586 to 4.7901] — LS Mean difference = LS Mean of Ampligen® - LS Mean of Placebo

7. Secondary Outcome: Change From Baseline to Week 6 and 13 in PROMIS Sleep Disturbance Score (T-Score)
Description: Change in mean sleep disturbance T-score as measured by PROMIS® (Patient-Reported Outcomes Measurement Information System) Sleep Disturbance - short form 4a that assesses self-perceived sleep quality. The lowest possible raw score is 4; the highest possible raw score is 20. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, with a standard deviation of 10 points. The lowest possible T-score is 32; the highest possible T-score is 73.3. A higher T-score represents more of the concept being measured, meaning the higher the T-Score, the worse the sleep disturbance of the individual. Scores <55 are within normal limits, 55-60 mild, 61-70 moderate, and >70 severe fatigue.
Time Frame: Baseline to Week 6 and 13
Population: All Modified Intent to Treat (mITT) Population
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Ampligen® /Rintatolimod | Placebo/Saline
Number analyzed (Participants) | 40 | 40
T-Score
  Baseline: number analyzed (Participants) | 37 | 39
  Baseline | 48.3 (7.99) | 48.4 (8.89)
  Change from baseline at Week6-V12: number analyzed (Participants) | 32 | 32
  Change from baseline at Week6-V12 | -10.9 (7.45) | -5.6 (9.21)
  change from baseline at Week13-V26: number analyzed (Participants) | 34 | 29
  change from baseline at Week13-V26 | -12.1 (7.95) | -10.7 (8.81)
Statistical Analysis 1: Comparison: Ampligen® /Rintatolimod vs Placebo/Saline; Test type: Superiority; p = 0.7823, ANCOVA; Mean Difference (Final Values) = -0.5161, 95% CI 2-sided [-4.2356 to 3.2035] — LS Mean difference = LS Mean of Ampligen® - LS Mean of Placebo

8. Other Pre Specified Outcome: Changes From Baseline in COVID-19-related Symptoms Using Symptom Burden Questionnaire for Long COVID (SBQ-LC) During the Course of the Treatment Phase.
Description: The SBQ-LC (Symptom Burden Questionnaire for Long COVID), which includes questions related to common COVID-19 symptoms, was assessed at baseline and at every odd-numbered visit from Visit 3 to Visit 25.
  Data at baseline and change from baseline at Week 12 (end of treatment) is reported.
  The converted scores reported for each symptom range from 0 to 100, with a higher score indicating worse symptom burden.
Time Frame: Baseline and the end of treatment phase at week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ampligen® /Rintatolimod | Placebo/Saline
Number analyzed (Participants) | 40 | 40
units on a scale
  Baseline : Breathing: number analyzed (Participants) | 37 | 39
  Baseline : Breathing | 21.5 (14.28) | 23.7 (16.97)
  Mean change from baseline at week12 : Breathing: number analyzed (Participants) | 33 | 28
  Mean change from baseline at week12 : Breathing | -19.2 (14.43) | -18.3 (12.70)
  Baseline : Circulation: number analyzed (Participants) | 37 | 39
  Baseline : Circulation | 9.4 (17.08) | 14.3 (20.94)
  Mean change from baseline at week12 : Circulation: number analyzed (Participants) | 33 | 28
  Mean change from baseline at week12 : Circulation | -6.4 (13.72) | -9.0 (12.61)
  Baseline : Ear, Nose, and Throat: number analyzed (Participants) | 37 | 39
  Baseline : Ear, Nose, and Throat | 9.5 (14.09) | 14.3 (17.50)
  Mean change from baseline at week12 : Ear, Nose, and Throat: number analyzed (Participants) | 33 | 28
  Mean change from baseline at week12 : Ear, Nose, and Throat | -5.4 (12.73) | -10.3 (14.26)
  Baseline: Eyes: number analyzed (Participants) | 37 | 39
  Baseline: Eyes | 8.8 (14.63) | 13.5 (19.25)
  change from baseline to week12 : Eyes: number analyzed (Participants) | 33 | 28
  change from baseline to week12 : Eyes | -3.9 (10.04) | -4.7 (10.64)
  Baseline Fatigue converted score: number analyzed (Participants) | 37 | 39
  Baseline Fatigue converted score | 28.1 (24.28) | 32.4 (27.87)
  change from baseline at week12 for fatigue score: number analyzed (Participants) | 33 | 28
  change from baseline at week12 for fatigue score | -22.0 (21.47) | -19.4 (23.06)
  Baseline: Female Repro.& Sex Health: number analyzed (Participants) | 17 | 16
  Baseline: Female Repro.& Sex Health | 4.6 (10.72) | 4.3 (6.77)
  change from baseline at week 12; Female Repro.& Sex Health: number analyzed (Participants) | 15 | 13
  change from baseline at week 12; Female Repro.& Sex Health | -2.8 (12.60) | -1.8 (6.85)
  Baseline: Impact on Daily Life Scale: number analyzed (Participants) | 37 | 39
  Baseline: Impact on Daily Life Scale | 13.7 (20.99) | 18.1 (24.01)
  Change from basline at week 12: Impact on Daily Life Scale: number analyzed (Participants) | 33 | 28
  Change from basline at week 12: Impact on Daily Life Scale | -9.2 (16.75) | -8.9 (15.18)
  Baseline:Male Repro.&Sex Health: number analyzed (Participants) | 20 | 23
  Baseline:Male Repro.&Sex Health | 12.2 (26.16) | 11.7 (21.29)
  change from baseline at week 12: Male Reproductive and Sexual Health: number analyzed (Participants) | 18 | 15
  change from baseline at week 12: Male Reproductive and Sexual Health | -3.2 (21.06) | -11.3 (20.47)
  Baseline: Memory,Thinking&Commun.: number analyzed (Participants) | 37 | 39
  Baseline: Memory,Thinking&Commun. | 13.7 (18.66) | 20.0 (23.64)
  Change from baseline to week 12; Memory,Thinking&Commun.: number analyzed (Participants) | 33 | 28
  Change from baseline to week 12; Memory,Thinking&Commun. | -7.5 (14.59) | -9.9 (20.23)
  Baseline: MentalHealth & Wellbeing: number analyzed (Participants) | 37 | 39
  Baseline: MentalHealth & Wellbeing | 28.2 (4.83) | 27.0 (7.22)
  Change from Baseline: MentalHealth & Wellbeing: number analyzed (Participants) | 33 | 28
  Change from Baseline: MentalHealth & Wellbeing | -17.1 (11.52) | -13.0 (16.48)
  Baseline: Movement: number analyzed (Participants) | 37 | 39
  Baseline: Movement | 10.8 (23.02) | 11.8 (25.39)
  Change from baseline at week 12: Movement: number analyzed (Participants) | 33 | 28
  Change from baseline at week 12: Movement | -5.5 (15.48) | -3.5 (8.68)
  Baseline: Muscle & Joints: number analyzed (Participants) | 37 | 39
  Baseline: Muscle & Joints | 11.5 (15.73) | 15.2 (22.09)
  change from baseline at week 12: Muscle & Joints: number analyzed (Participants) | 33 | 28
  change from baseline at week 12: Muscle & Joints | -7.3 (11.77) | -6.1 (12.09)
  Baseline: Other Symptoms: number analyzed (Participants) | 37 | 39
  Baseline: Other Symptoms | 10.9 (13.75) | 13.2 (15.64)
  Change from baseline at week 12: Other Symptoms: number analyzed (Participants) | 33 | 28
  Change from baseline at week 12: Other Symptoms | -8.1 (11.29) | -7.9 (11.72)
  Baseline: Pain Scale: number analyzed (Participants) | 37 | 39
  Baseline: Pain Scale | 5.5 (9.45) | 7.4 (14.53)
  Change from Baseline at week12: Pain Scale: number analyzed (Participants) | 33 | 28
  Change from Baseline at week12: Pain Scale | -3.2 (8.94) | -4.1 (8.13)
  Baseline: Skin & Hair: number analyzed (Participants) | 37 | 39
  Baseline: Skin & Hair | 10.9 (14.32) | 12.2 (20.13)
  Change from baseline at week12: Skin & Hair: number analyzed (Participants) | 33 | 28
  Change from baseline at week12: Skin & Hair | -8.2 (13.05) | -3.8 (9.53)
  Baseline: Sleep Scale: number analyzed (Participants) | 37 | 39
  Baseline: Sleep Scale | 31.0 (31.68) | 35.1 (30.53)
  Change from Baseline at week12: Sleep Scale: number analyzed (Participants) | 33 | 28
  Change from Baseline at week12: Sleep Scale | -18.4 (30.99) | -23.8 (28.27)
  Baseline: Stomach & Digestion: number analyzed (Participants) | 37 | 39
  Baseline: Stomach & Digestion | 6.6 (12.71) | 10.1 (14.83)
  Change from Baseline: Stomach & Digestion: number analyzed (Participants) | 33 | 28
  Change from Baseline: Stomach & Digestion | -4.0 (12.21) | -4.7 (9.03)

9. Other Pre Specified Outcome: Change From Baseline in Cognitive Function as Measured by Montreal Cognitive Assessment (MoCA) at Weeks 4, 8, and 13 During the Treatment Phase
Description: The change from baseline in Montreal Cognitive Assessment (MoCA) at week 4, 8, and 13 is presented and summarized descriptively by treatment group. Higher scores indicate better cognitive function; total scores equal to or higher than 26 are considered normal.
  Montreal Cognitive Assessment range is from 0-30, with a score of 26 or higher indicating normal cognitive function. 18-25 indicates mild cognitive impairment; 10-17 indicates moderate cognitive impairment; less than 10 indicates severe cognitive impairment.
Time Frame: Baseline to weeks 4, 8 and 13 during treatment phase
Population: The Modified Intent-to-Treat (mITT) population is defined as the set of subjects whohave received at least one dose of study treatment (Ampligen® or placebo).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ampligen® /Rintatolimod | Placebo/Saline
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline: number analyzed (Participants) | 39 | 40
  Baseline | 27.7 (2.04) | 28.1 (2.06)
  change from baseline at Week 4 - V8: number analyzed (Participants) | 35 | 34
  change from baseline at Week 4 - V8 | -0.6 (3.61) | -0.1 (2.8)
  change from baseline at Week 8 - v16: number analyzed (Participants) | 35 | 33
  change from baseline at Week 8 - v16 | -0.1 (2.75) | -0.2 (3.14)
  change from baseline at Week 13 - V26: number analyzed (Participants) | 36 | 30
  change from baseline at Week 13 - V26 | 0.8 (2.26) | 0.5 (2.11)
Statistical Analysis 1: Comparison: Ampligen® /Rintatolimod vs Placebo/Saline; Test type: Superiority; p = 0.5185, ANCOVA; Mean Difference (Final Values) = 0.2779, 95% CI 2-sided [-0.5775 to 1.1333] — LS Mean difference = LS Mean of Ampligen® - LS Mean of Placebo

10. Other Pre Specified Outcome: Hospitalizations
Description: Number of subjects with hospitalization during treatment phase up to week 12.
Time Frame: During the treatment phase up to 12 weeks
Population: all Modified Intent-to-Treat population subjects
Measure: Number; unit: participants
Groups:
- Experimental: Ampligen / Rintatolimod: Subjects received rintatolimod (intravenous [IV]), up to 400 mg twice weekly for 12 weeks.
- Placebo Comparator: Placebo / Saline: Subjects received placebo / normal saline (intravenous [IV]), up to 160 mL twice weekly for 12 weeks.
Arm/Group | Experimental: Ampligen / Rintatolimod | Placebo Comparator: Placebo / Saline
Number analyzed (Participants) | 40 | 40
participants | 0 | 0
Statistical Analysis 1: Comparison: Experimental: Ampligen / Rintatolimod vs Placebo Comparator: Placebo / Saline; Test type: Other; No patients were hospitalized

11. Other Pre Specified Outcome: Duration of Hospitalizations
Description: Duration (days) of hospitalization during the treatment phase up to week 12.
Time Frame: During the treatment phase up to 12 weeks
Population: No patients were hospitalized.
Arm/Group | Ampligen / Rintatolimod | Placebo / Saline
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Evaluation of Lymphocyte Profile by Flow Cytometry in Patients With Post-COVID-19 Conditions - Absolute Value of CD3+
Description: A blood sample was collected at V2 (pre-dose), V12 (pre-dose), and V26 (Follow-up 1) for research purposes to conduct exploratory analyses of lymphocyte profile by flow cytometry. The absolute values and change from baseline data for CD3+ were evaluated.
Time Frame: Baseline to week 6 and 13
Population: all Modified Intent-to-Treat population subjects
Measure: Mean (Standard Deviation); unit: CD3+ cells/μL
Arm/Group | Ampligen® /Rintatolimod | Placebo/Saline
Number analyzed (Participants) | 40 | 40
CD3+ cells/μL
  Baseline: number analyzed (Participants) | 25 | 20
  Baseline | 1598.4 (573.79) | 1739.4 (637.33)
  Change from Baseline to Week6-V12: number analyzed (Participants) | 19 | 17
  Change from Baseline to Week6-V12 | -54.1 (756.11) | -71.8 (389.79)
  Change from Baseline to Week13-V26: number analyzed (Participants) | 16 | 14
  Change from Baseline to Week13-V26 | 65.8 (532.92) | -196.3 (324.0)
Statistical Analysis 1: Comparison: Ampligen® /Rintatolimod vs Placebo/Saline; Test type: Superiority; p = 0.2175, ANCOVA; Mean Difference (Final Values) = 169.3890, 95% CI 2-sided [-105.892 to 444.6702] — LS Mean difference = LS Mean of Ampligen® - LS Mean of Placebo; LS Mean difference = LS Mean of Ampligen® - LS Mean of Placebo

13. Other Pre Specified Outcome: Evaluation of Lymphocyte Profile by Flow Cytometry in Patients With Post-COVID-19 Conditions - Absolute Value of CD3-CD56+ Natural Kill
Description: A blood sample was collected at V2 (pre-dose), V12 (pre-dose), and V26 (Follow-up 1) for research purposes to conduct exploratory analyses of lymphocyte profile by flow cytometry. The absolute values and change from baseline data for CD3-CD56+ natural killers (NK+) were evaluated.
Time Frame: Baseline to week 6 and 13
Population: all Modified Intent-to-Treat population subjects
Measure: Mean (Standard Deviation); unit: CD3-CD56+ Natural Killer cells/μL
Arm/Group | Ampligen® /Rintatolimod | Placebo/Saline
Number analyzed (Participants) | 40 | 40
CD3-CD56+ Natural Killer cells/μL
  Baseline: number analyzed (Participants) | 33 | 31
  Baseline | 252.5 (120.11) | 235.1 (113.55)
  Change from Baseline to Week6-V12: number analyzed (Participants) | 26 | 28
  Change from Baseline to Week6-V12 | -27.2 (137.66) | -28.3 (116.7)
  Change from Baseline to Week13-V26: number analyzed (Participants) | 26 | 22
  Change from Baseline to Week13-V26 | -27.9 (75.45) | 25.4 (215.0)
Statistical Analysis 1: Comparison: Ampligen® /Rintatolimod vs Placebo/Saline; Test type: Superiority; p = 0.2086, ANCOVA; Mean Difference (Final Values) = -56.9984, 95% CI 2-sided [-147.021 to 33.0241] — LS Mean difference = LS Mean of Ampligen® - LS Mean of Placebo; LS Mean difference = LS Mean of Ampligen® - LS Mean of Placebo

14. Other Pre Specified Outcome: Evaluation of Lymphocyte Profile by Flow Cytometry in Patients With Post-COVID-19 Conditions - CD4:CD8 Ratio
Description: A blood sample was collected at V2 (pre-dose), V12 (pre-dose), and V26 (Follow-up 1) for research purposes to conduct exploratory analyses of lymphocyte profile by flow cytometry. The absolute values and change from baseline data for CD4:CD8 ratio were evaluated.
Time Frame: Baseline to week 6 and 13
Population: all Modified Intent-to-Treat population subjects
Measure: Mean (Standard Deviation); unit: CD4:CD8 Ratio
Arm/Group | Ampligen® /Rintatolimod | Placebo/Saline
Number analyzed (Participants) | 40 | 40
CD4:CD8 Ratio
  Baseline: number analyzed (Participants) | 39 | 35
  Baseline | 1.7 (0.7) | 1.6 (0.58)
  Change from Baseline to Week6-V12: number analyzed (Participants) | 33 | 29
  Change from Baseline to Week6-V12 | 0.0 (0.36) | 0.0 (0.28)
  Change from Baseline to Week13-V26: number analyzed (Participants) | 35 | 25
  Change from Baseline to Week13-V26 | 0.2 (0.48) | 0.0 (0.19)
Statistical Analysis 1: Comparison: Ampligen® /Rintatolimod vs Placebo/Saline; Test type: Superiority; p = 0.0975, ANCOVA; Mean Difference (Final Values) = 0.1733, 95% CI 2-sided [-0.0327 to 0.3792] — LS Mean difference = LS Mean of Ampligen® - LS Mean of Placebo; LS Mean difference = LS Mean of Ampligen® - LS Mean of Placebo

15. Other Pre Specified Outcome: Identification and Evaluation of Plasma Protein Biomarkers in Patients With Post-COVID-19 Conditions
Description: A blood sample was collected at V2 (pre-dose) and V26 (Follow-up 1) for research purposes to conduct exploratory analyses of protein biomarkers.
Time Frame: Baseline and week 13
Reporting Status: Not Posted

16. Post Hoc Outcome: Change From Baseline to Week 6 and Week 13 in Distance Traveled During 6-minute Walk Test (6MWT) - Subjects Walking ≥205 Meters at Baseline
Description: as for outcome 4
Time Frame: Baseline to week 6 and week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Ampligen® /Rintatolimod | Placebo/Saline
Number analyzed (Participants) | 35 | 35
Meters
  Baseline | 337.3 (63.79) | 328.9 (74.3)
  Change from baseline at week6-V12: number analyzed (Participants) | 32 | 29
  Change from baseline at week6-V12 | -21.8 (72.65) | -9.3 (89.39)
  Change from baseline at week13-V26: number analyzed (Participants) | 32 | 25
  Change from baseline at week13-V26 | 81.3 (114.37) | 64.9 (98.2)
Statistical Analysis 1: Comparison: Ampligen® /Rintatolimod vs Placebo/Saline; Test type: Superiority; p = 0.4545, ANCOVA; Mean Difference (Final Values) = 20.7131, 95% CI 2-sided [-34.4079 to 75.8341] — LS Mean Difference - LS Mean of Ampligen® - LS Mean of Placebo

17. Post Hoc Outcome: Change From Baseline to Week 6 and Week 13 in Distance Traveled During 6-minute Walk Test (6MWT) - Subjects Walking <205 Meters at Baseline
Description: as for outcome 4
Time Frame: Baseline to week 6 and week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Ampligen® /Rintatolimod | Placebo/Saline
Number analyzed (Participants) | 5 | 5
Meters
  Baseline | 180.0 (22.45) | 194.4 (15.65)
  Change from baseline at week6-V12 | 123.6 (101.96) | 63.0 (43.06)
  Change from baseline at week13-V26 | 139.2 (18.2) | 91.2 (27.63)
Statistical Analysis 1: Comparison: Ampligen® /Rintatolimod vs Placebo/Saline; Test type: Superiority; p = 0.0333, ANCOVA; Mean Difference (Final Values) = 44.1231, 95% CI 2-sided [4.6338 to 83.6123] — LS Mean Difference - LS Mean of Ampligen® - LS Mean of Placebo

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: AEs reported through direct questioning and subject reports. An AE is defined as any unfavorable or unintended sign, symptom, or disease that occurred or was reported by the patient to have occurred, or the worsening of a pre-existing condition. Any abnormality in physical examination findings or laboratory results that the investigator believes is clinically significant (CS) to the research subject and that occurred after initiation of the first study treatment were reported as AEs.
Arm/Group | Ampligen / Rintatolimod | Placebo / Saline
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 10/40 | 4/40
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ampligen / Rintatolimod (N=40) | Placebo / Saline (N=40)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Paraesthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Injection site phlebitis (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study didn't aim to establish statistical significance of Ampligen® over placebo. Sample size of 80 subjects was based on clinical judgement and no statistical power calculation was used. Fatigue itself, along with cognitive function and sleep, is a multidimensional measure and can be influenced by many factors beyond study treatment, such as general health status, physical activity, etc. Placebo effect is a known challenge, particularly when using patient-reported outcomes as study endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT05592418/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT05592418/SAP_001.pdf